CLINICAL TRIAL: NCT00967759
Title: A Double Blind, Randomized, Multicenter Phase III Study Comparing 3 Formulations: Dose Fixed Combination of Bronpheniramine and Fenilefrine, Bronpheniramine Isolated and Fenilefrine Isolated, to Evaluate the Efficacy and Safety of the Treatment of the Inflammatory Symptoms of Upper Respiratory Tract, in Children Between 2 and 6 Years Old.
Brief Title: Study Comparing 3 Formulations to Evaluate the Efficacy and Safety of the Inflammatory Symptoms of the Upper Respiratory Tract, in Children Between 2 and 6 Years Old
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was designed again in compliance with the regulatory agency.
Sponsor: Ache Laboratorios Farmaceuticos S.A. (Industry)
Responsible Party: Carla Rosana Goulart Silva Peron, MD, Ache Laboratorios Farmaceuticos S.A.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ACH-DCN-03(05/08)
Record Dates: First submitted 2009-08-26; First posted 2009-08-28 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Common Cold
Keywords: common cold; treatment; inflammatory symptoms of superior air passages affection
MeSH Terms: conditions — Common Cold

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Decongex Plus (Experimental)
  Interventions: Drug: Bronpheniramine and fenilefrine (Decongex Plus)
- Bronpheniramine isolated (Active Comparator)
  Interventions: Drug: Bronpheniramine isolated
- Fenilefrine isolated (Active Comparator)
  Interventions: Drug: Fenilefrine isolated

INTERVENTIONS:
Drug: Bronpheniramine and fenilefrine (Decongex Plus) — Oral Solution: Bronpheniramine (2mg/ml) and fenilefrine (2,5mg/ml) 2 drops/kg/day divided into 3 doses; maximum of 60 drops/day QID, during 5 days.
  Arms: Decongex Plus
Drug: Bronpheniramine isolated — Oral Solution: Bronpheniramine (2mg/ml) 2 drops/kg/day divided into 3 doses; maximum of 60 drops/day QID, during 5 days.
  Arms: Bronpheniramine isolated
Drug: Fenilefrine isolated — Oral Solution: Fenilefrine (2,5mg/ml) 2 drops/kg/day divided into 3 doses; maximum of 60 drops/day QID, during 5 days.
  Arms: Fenilefrine isolated

SUMMARY:
The primary outcome of this study is to evaluate the clinical efficacy of the dose fixed combination and each drug, that composes it, isolated, regarding the respiratory symptoms improvement in superior air passages acute affection in children between 2 and 6 years old.

ELIGIBILITY:
Inclusion Criteria:

1. Patients between 2 and 6 years old, according to dosage information provided in the product package insert.
2. Patient with a relative available for observation of symptoms during the night.
3. Patients with acute symptoms of air passages jeopardizing, initiated, at least, 24 hours before patient inclusion in this protocol and, at most, in the 3 days before patient inclusion.
4. Patients facing at least a 7 points score in the addition of general symptoms (rhinorrhea, sneeze, itching, nose obstruction and coughing).
5. At least two symptoms must be moderated in scale, for specific evaluation.
6. Presence of fluid and/or sputum verified through a rhinoscopy.

Exclusion Criteria:

1. Children younger than 2 years old or a weight and/or height percentual inferior to 10.
2. Children with corporal weight superior to 30Kg.
3. Suggestive signs of superior air passages bacterial infection to the rhinoscopy, otoscopy and oropharingoscopy.
4. Chronic oral breath with a 6 months history.
5. Presence of degree II and III of nasal septal deviation (in any region and in any nasal fossa) and/or presence of nasal polyp or other conditions that determine nasal obstruction.
6. Patients in a chronic medication treatment for allergy.
7. Patients with an asthma clinical history confirmed (diagnosed).
8. Personal preceding of nasal surgery that in the opinion of the investigator can influence in the resistance to the air nose flow.
9. Children older than 5 years old that are not registered in the school.
10. Children that don´t have vaccination notebook.
11. Patient that had used prohibited medication, during the established period before V0 - Randomization Visit (See Picture 1).
12. Hypersensitive history to the study drug or its components.
13. Patient that have participated in, during the last 12 months, study protocols (according to Resolution 251, dated of August, 7th 1997, item III, sub-item J, "Investigator Responsibility", its recommended that the same person does not be subject of a clinical study in a new project before have elapsed 1(one) year from previous study participation, unless there is a direct benefit to the study patient).
14. Relatives of sponsor´s or study site´s employee.
15. Patients with gastroesofagic reflux disease.
16. Presence of psychiatry diseases.
17. Presence of mental disorder of any etiology.
18. Renal and hepatic insufficiency.
19. Patient with current evidence of clinically significant diseases, of origin: hematopoietic, gastrointestinal, cardiovascular, hepatic, renal, neurological, endocrinological, psychiatric, self immune, pulmonary, or other that preclude, according to the investigator criteria, the subject participation.
20. Patients with genetic diseases.
21. Any finding of clinical observation (anamneses and physical evaluation) that be understood by the investigator as risk to the patient participation in the study.
22. Any finding of lab result that the investigator judges as a risk to the patient, considering the participation in the study.
23. Patients with AST and ALT levels higher than 20% related to the upper normal limits; total bilirubins with an increase of 10% related to the upper normal limits; fasting serum/blood glucose >99mg/dl or postprandial serum/blood glucose >140mg/dl; Hb <10g/dl ou Hb >15 g/dl; serum creatinine with levels over than 10% of upper limit; serum potassium under 3,5 mEq/L, or upper 5,1 mEq/L; serum sodium under 136 mEq/L, or upper 145 mEq/L.
24. Presence of hematogenous or meliceric, purulent or mucus purulent secretion, bulging or malformation (leporine lips and nasolabial fissure surgically corrected or not) in the region of the nasal vestibule.

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Evaluate the clinical efficacy of the dose fixed combination and each drug, that compose it, isolated, regarding the respiratory symptoms improvement in superior air passages acute affection in children between 2 and 6 years old. | 04/2010

SECONDARY OUTCOMES:
Patient adherence to the treatment. | 04/2010
Use of co intervention for symptom relief during treatment | Assessed during the treatment in the diary and questioned by the Investigator at the visits
Evaluate the intensity of the symptoms during the treatment | Assessed during the treatment
Adverse effect appearance during the study and tolerability | Assessed during the treatment and at the final visit

CONTACTS AND LOCATIONS:
Overall Officials: Luc Weckx, MD, Principal Investigator — Federal University of São Paulo; Fabio Castro, MD, Principal Investigator — Instituto de Medicina Avançada; Flavio Sano, MD, Principal Investigator — Hospital Beneficência Nipo Brasileiro
Locations (1):
- UNIFESP, São Paulo, São Paulo, Brazil